CLINICAL TRIAL: NCT03173781
Title: Effects of Droxidopa When Measuring Gait Speed, Kyphosis, and Functional Reach in Parkinson's Disease
Acronym: droxidopa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado Springs Neurological Associates (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSNA001
Record Dates: First submitted 2016-08-10; First posted 2017-06-02 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Droxidopa; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- droxidopa (Experimental): Droxidopa will be supplied in 100 and 200 mg pill sizes. The subject should administer the three doses 4 hours apart with the last dose prior to 4:00 pm (example: 8:00 am, 12:00 pm, and 4:00 pm). The proposed dosing is 100mg TID at baseline, then titrate slowly up to 600 mg TID. During titration, droxidopa or placebo, initiated at 100 mg TID was titrated upward in 100-mg TID increments every 48 hours until the subject:
  1. Reaches the maximum permitted dosage of 600 mg TID;
  2. Has a systolic blood pressure≥160mmHg or diastolic blood pressure ≥100mmHg after 10 minutes supine on 3 consecutive measurements; or
  3. Experiences intolerable adverse events (AEs).
  Interventions: Drug: droxidopa
- placebo (Placebo Comparator): sugar pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: droxidopa — medication
  Other Names: Northera
  Arms: droxidopa
Drug: Placebo — medication
  Other Names: sugar pill
  Arms: placebo

SUMMARY:
The purpose of this study is to determine if droxidopa reduces fall risk by improving gait speed, kyphosis, and functional reach in individuals with Parkinson's disease.

DETAILED DESCRIPTION:
Gait disorders and balance impairments are one of the most incapacitating symptoms of Parkinson's disease (PD). Gait impairment in Parkinson's disease exists despite the use of dopinergic therapy. Motor phenotype associated with postural instability and ambulatory dysfunction is related to greater risk of motor decline and may be influenced by non-dopinergic pathology (Galna et al., 2015). Galna et al. (2015) conducted a study to document the progression of gait impairment over 18 months in individuals with Parkinson's disease with regard to phenotype and medication. Gait characteristics were measured in 121 PD and 184 controls, and 18 months later in 108 PD participants (Galna, 2015). Sixteen gait characteristics were examined with respect to five broad domains for PD and motor phenotype. Correlations between change in levodopa (l-dopa) equivalent daily dose and gait were used to identify dopa-responsive and nonresponsive characteristics (Galna, 2015). Pace and rhythm deteriorated over 18 months in people with PD, with other gait domains remaining stable. People with a postural instability and gait difficulty phenotype had more impaired gait at baseline compared with a tremor-dominant phenotype, which was most evident in temporal characteristics (Galna, 2015). In contrast, pace and variability deteriorated over the subsequent 18 months in the tremor-dominant phenotype only (Galna, 2015). Weak but statistically significant correlations were found between increased l-dopa medication and less deterioration in pace and asymmetry. Significant gait impairment is evident in very early disease despite optimal medication (Galna, 2015).

For people with Parkinson's disease, there are fall risk factors specific to PD. These include changes in posture, postural instability, freezing of gait, dyskinesias, gait changes, medication side effects, and decreased ability to react automatically to a loss of balance. Health and cognitive factors such as cognitive decline and depression can also greatly increase the risk of falling. Contreras and Grandas (2012) conducted a study in Spain that included 160 people with Parkinson's disease who were being seen at a movement disorders clinic in Madrid. It was found that that fallers were older and had longer disease duration (Contreras & Grandas, 2012). Subjects also had increased disease severity according to the UPDRS (part III) and the Hoehn and Yahr scale, and lower scores on the Schwab and England ADL test (Contreras & Grandas, 2012). In addition, fallers scored worse in the Mini-Mental State Examination and experienced a higher frequency of motor fluctuations, dyskinesia, and freezing of gait (Contreras & Grandas, 2012).

Among people with PD, recurrent falls are more frequent, with one study reporting that more than 50% of the study participants fell recurrently. In another study involving a survey of 100 people with PD, 13% reported falling more than once a week, with most of these people falling multiple times a day (Allen et al., 2013). Several risk factors for falls have been found to be more strongly associated with recurrent falls than single falls. Some of these factors are potentially modifiable, including cognitive impairment, freezing of gait, fear of falling, reduced mobility, reduced physical activity, and balance impairments (Allen et al., 2013). There is substantial variability in the falling rates reported in various studies, with the proportion of fallers (single and recurrent) ranging from 35% to 95%. Differences in the method of monitoring falls could contribute to this variability (Allen et al., 2013). Despite the fact that recurrent falls are a substantial problem for people with PD, the scope of, and risk factors for, recurrent falls in PD are not clearly understood (Allen et al., 2013).

Elbers et al. (2012) investigated the predictive value of gait speed for community walking in Parkinson's disease. A total of 153 patients with Parkinson's disease were included in this study. Community walking was evaluated using the mobility domain of the Nottingham Extended Activities of Daily Living Index (NEAI). Patients who scored 3 points on item 1 ("Did you walk around outside?") and item 5 ("Did you cross roads?") were considered community walkers (Elbers et al., 2012). Gait speed was measured with the 6-m or 10-m timed walking test. Age, gender, marital status, disease duration, disease severity, motor impairment, balance, freezing of gait, fear of falling, previous falls, cognitive function, executive function, fatigue, anxiety and depression were investigated for their contribution to the multivariate model (Elbers et al., 2012). Results indicated seventy patients (46%) were classified as community walkers. A gait speed of 0.88 m/s correctly predicted 70% of patients as community walkers (Elbers et al., 2012). A multivariate model, including gait speed and fear of falling, correctly predicted 78% of patients as community walkers (Elbers et al., 2012). Elbers et al. concluded timed walking tests are valid measurements to predict community walking in Parkinson's disease. However, evaluation of community walking should include an assessment of fear of falling.

Combs et al. (2013) conducted a study to determine test-retest reliability and responsiveness of short-distance walking speed tests for persons with Parkinson disease (PD). Discriminant and convergent validity of walking speed tests were also examined. Eighty-eight participants with PD (mean age, 66 years) with mild to moderate severity (stages 1-4 on the Hoehn and Yahr Scale) were tested on medications. Measures of activity included the comfortable and fast 10-m walk tests (CWT, FWT), 6-min walk test (6MWT), mini balance evaluations systems test (mini-BEST Test), fear of falling (FoF), and the Activity-Specific Balance Confidence Scale (ABC). The mobility subsection of the PD quality of life-39 (PDQ39-M) served as a participation-based measure (Combs et al., 2013). Results indicated test-retest reliability was high for both walking speed measures (CWT, ICC(2,1) = 0.98; FWT, ICC(2,1) = 0.99) (Combs et al., 2013). Minimal detectable change (MDC(95)) for the CWT and FWT was 0.09 m/s and 0.13 m/s respectively (Combs et al., 2013). Participants at Hoehn & Yahr levels 3/4 demonstrated significantly slower walking speed with the CWT and FWT than participants at Hoehn & Yahr levels 1 and 2 (P < .01). The CWT and FWT were both significantly (P ≤ .002) correlated with all activity and participation-based measures (Combs et al., 2013). In conclusion, short-distance walking speed tests are clinically useful measures for persons with PD (Combs et al., 2013). The CWT and FWT are highly reliable and responsive to change in persons with PD (Combs et al., 2013). Short distance walking speed can be used to discriminate differences in gait function between persons with mild and moderate PD severity (Combs et al., 2013). The CWT and FWT had moderate to strong associations with other activity and participation based measures demonstrating convergent validity (Combs et al., 2013).

Patients with Parkinson's disease (PD) or atypical parkinsonism often present with abnormal posture. A retrospective observational study conducted by Doherty et al. (2011) showed that a third of patients with PD had a deformity of their limbs, neck, or trunk. The most recognized type of deformity is the classic stooped simian appearance, with flexion of the hips and knees, and rounding of the shoulders (Doherty et al., 2011). Severe postural deformities include kyphosis, camptocormia, antecollis, Pisa syndrome, and scoliosis. The underlying pathophysiology of these deformities is largely unknown, and their management remains difficult (Doherty et al., 2011).

Thoracic hyperkyphosis is one of the most common postural abnormalities. It is defined as increased thoracic curvature in the sagittal plan of the vertebral column. Normal kyphosis may range from 20º to 50º according to Cobb's radiographic method. The radiographic method is the most popular kyphosis measuring method, but because it is an expensive method and it exposes the individual to radiation, it is not the most appropriate method for periodic patient follow-up. Routine clinical examinations such as physiotherapeutic evaluation of thoracic kyphosis need to be valid, reliable, sensitive, practical and cheap.

A study by Teixeira and Carvalho (2007) assessed the reliability and validity of thoracic kyphosis measurements using the flexicurve method. A cross-sectional study analyzed the thoracic kyphosis of 56 people from sagittal radiography of the thoracic column using Cobb's method and by means of the flexicurve method, by two evaluators. Results indicated he intra-class correlation coefficient (ICC) between the measurements from the Cobb and flexicurve methods was 0.906 (Teixeira & Carvalho, 2007). For diagnosing thoracic hyperkyphosis, the sensitivity was 85% and the specificity was 97% (Teixeira & Carvalho, 2007). In conclusion, the flexicurve method was shown to be a suitable quantitative clinical method for measuring the curvature of thoracic kyphosis (Teixeira & Carvalho, 2007).

The Get Up and Go test, the predecessor of the Timed Up and Go test (TUG), was developed by Mathias and Nayak as a tool to screen for balance problems, primarily in the frail elderly. The test measures how long it takes for a person to rise from a chair, walk 3 meters (about 10 feet) to a line on the floor, and return to the chair. The test correlates well with the Berg Balance Scale, the Barthel Index of activities of daily living, and gait speed tests. The Timed Up and Go modified the earlier version of the test by adding a timing component. An adult who is independent in balance and mobility can perform the TUG in less than 10 seconds (Shumway-Cook & Woollacott, 2007). In a study of older adults with a range of neurologic pathologies, people taking 30 seconds or more to complete the TUG were more likely to need an assistive device, walk too slowly for community ambulation, and score lower on the Berg Balance scale. In contrast, a person completing the test in less than 20 seconds was more likely to be independent in daily living activities, score higher on the Berg Balance scale, and walk at a speed sufficient for community mobility (Podsiadlo & Richardson, 1991). Shumway-Cook and Woollacott (2012) noted that the TUG can be used to predict the risk of falls in older adults. In a study, 30 community-dwelling frail elderly adults were tested using the TUG, and researchers found that those taking longer than 14 seconds to complete the task were at high risk for falls. In the same study, the TUG was modified by adding a cognitive task (counting backward by threes) and a manual task (carrying a full cup of water). The addition of a secondary task increased the time need to complete the TUG by 22% to 25% (Shumway-Cook & Woollacott, 2012).

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

1. 18 years of age or older.
2. Clinical diagnosis of Parkinson's disease.
3. Stable dose of current Parkinson's disease medication(s) for the past 2 weeks.
4. Stable deep brain stimulator settings for the past 2 weeks.
5. Provide written informed consent to participate in the study.

Exclusion Criteria:

1. Concomitant use of vasoconstricting agents for the purpose of increasing blood pressure.

   Patients taking vasoconstricting agents such as ephedrine, dihydroergotamine, or midodrine must stop taking these drugs at least 2 days prior to baseline and throughout the duration of the study.
2. Concomitant use of the following medications:
3. Anti-hypertensive medication for the treatment of essential hypertension
4. Vasoconstricting agents such as ephedrine, dihydroergotamine, or midodrine. Concomitant treatment for symptomatic NOH (with the exception of vasoconstricting agents) will be permitted during the study. This includes fludrocortisone, which is permitted during the study. Medications for the treatment of PD will be permitted during the study.
5. Sumatriptan-like drugs, (for example, naratriptan, zolmitriptan, rizatriptan)
6. Cyclopropane or halothane, or other halogen-containing inhalational anesthetics
7. Catecholamine-containing preparations (e.g. isoprenaline)
8. Non-selective monoamine oxidase inhibitors (MAOIs)
9. Ergotamine derivatives (except if anti-Parkinsonian medication)
10. Any investigational medication.
11. Uncontrolled depression.
12. Prior history of neuroleptic malignant syndrome.
13. History of suicide attempt within the previous 2 years.
14. Known or suspected alcohol or substance abuse within the past 12 months (DSM-IV definition of alcohol or substance abuse).
15. Women who are pregnant or breastfeeding.
16. Women of child bearing potential (WOCP) who are not using at least one method of contraception with their partner.
17. Male patients who are sexually active with a woman of child bearing potential (WOCP) and not using at least one method of contraception.
18. Untreated closed angle glaucoma, or treated closed angle glaucoma that, in the opinion of an ophthalmologist, might result in an increased risk to the patient.
19. Sustained severe hypertension (BP ≥ 180 mmHg systolic or ≥ 110 mmHg diastolic in the seated or supine position which is observed in 3 consecutive measurements over an hour).
20. Any significant uncontrolled cardiac arrhythmia.
21. History of myocardial infarction, within the past 2 years.
22. Current unstable angina.
23. Congestive heart failure (NYHA Class 3 or 4).
24. Diabetic autonomic neuropathy.
25. History of cancer within the past 2 years other than a successfully treated, non-metastatic cutaneous squamous cell or basal cell carcinoma or cervical cancer in situ.
26. Gastrointestinal condition, which in the Investigator's judgment, may affect the absorption of study drug (e.g. ulcerative colitis, gastric bypass).
27. Any major surgical procedure within 30 days of the baseline visit
28. Previous or current treatment with droxidopa.
29. Current participation in individual physical therapy, specifically for balance or gait.
30. Any condition or laboratory test result, which in the Investigator's judgment, might result in an increased risk to the patient, or would affect their participation in the study.
31. Additionally the Investigator has the ability to exclude a patient if for any reason they feel the subject is not a good candidate for the study or will not be able to follow study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-04; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of droxidopa when measuring walking speed using the 10 meter walk test . | 24 months
  10 meter walk test
  * Subject walks without assistance 10 meters (32.8 feet).
  * Assistive devices can be used but should be kept consistent and documented from test to test.
  * If physical assistance is required to walk, this should not be performed
  * Collect three trials and calculate the average of the three trials
  * Individuals are permitted to use the assistive device they typically use in the community, but without the assistance of another person.
Evaluate the efficacy of droxidopa when measuring walking speed using Dual Task Timed Up and Go test | 24 months
  * Subjects are given verbal instructions to stand up from a chair, walk 3 meters as quickly and safely as possible, cross a line marked on the floor, turn around, walk back, and sit down.
  * In the TUG (Cognitive), individuals were asked to complete the test while counting backward by threes from a randomly selected number between 20 and 100.

SECONDARY OUTCOMES:
Evaluate the efficacy of droxidopa when measuring degree of thoracic curvature using the Flexicurve rule | 24 months
  Flexi-curve measurement
  * Instruct subject to "stand in your usual best posture"
  * Identify C7 spinous process.
  * Identify the L-S interspace.
  * Mark each landmark (C7 process and L-S space) with a single horizontal grease pencil line.
  * Make sure the patient is standing in their usual best posture so that the marks are in the correct place during measurement using flexi-curve ruler.
Evaluate the efficacy of droxidopa when measuring fall risk using the Forward Functional Reach test. | 24 months
  Forward Functional Reach test
  * Using a yardstick mounted on the wall at shoulder height, ask the subject to position body close to, but not touching the wall with arm outstretched and hand fisted. Take note of the starting position by determining what number the MCP joints line up with on the rule.
  * Have the subject reach as far forward as possible in a plane parallel with the measuring device.
  * Instruct subject to "Reach as far forward as you can go without taking a step." Subjects are free to use various reaching strategies.
  * Take note of the end position of the MCP joints against the ruler, and record the difference between the starting and end position numbers.
  * If the feet move, that trial must be discarded and repeated.

CONTACTS AND LOCATIONS:
Overall Officials: Christen Kutz, PhD, PA-C, Study Director — Colorado Springs Neurological Associates
Locations (1):
- Colorado Springs Neurological Associates, Colorado Springs, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
movement disorder meeting/poster/paper